CLINICAL TRIAL: NCT01680419
Title: Mission Reconnect: Promoting Resilience and Reintegration of Post-Deployment Veterans and Their Families
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Collinge and Associates, Inc. (Other)
Responsible Party: Principal Investigator, William Collinge, PhD, President, Collinge and Associates, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R44MH088063-02 (NIH)
Record Dates: First submitted 2012-08-31; First posted 2012-09-07 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Stress; Depression; PTSD; Sleep; Compassion
Keywords: Veterans; Reintegration; Resilience; Marital; Spouse; Behavioral intervention; PTSD; Integrative therapies; Complementary therapies; Massage; Meditation; Mindfulness; Compassion; Mental health
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mission Reconnect only (Experimental): Autonomous use of the Mission Reconnect multimedia instructional program at home.
  Interventions: Behavioral: Mission Reconnect
- PREP only (Active Comparator): Participation in a standard PREP for Strong Bonds weekend retreat program.
  Interventions: Behavioral: PREP
- PREP plus Mission Reconnect (Active Comparator): Participation in a standard PREP for Strong Bonds weekend retreat followed by autonomous use of the Mission Reconnect multimedia instructional program at home.
  Interventions: Behavioral: Mission Reconnect; Behavioral: PREP
- Wait-list control (No Intervention): No intervention, followed by delivery of the Mission Reconnect multimedia program materials for home use after the end of the study period.

INTERVENTIONS:
Behavioral: Mission Reconnect — Multimedia package (audio, video, and print, web-based and downloadable to mobile devices) comprising an integrated program of (1) guided mind/body stress reduction and relaxation practices, (2) contemplative practices to engender and support appreciation, empathy and forgiveness for oneself and one's loved ones, and (3) video instruction in use of simple massage techniques with a partner for connection and stress reduction.
  Arms: Mission Reconnect only; PREP plus Mission Reconnect
Behavioral: PREP — The Army's "PREP for Strong Bonds" program offers retreats for partnered soldiers to support reintegration and healthy relationships. PREP (Prevention and Relationship Enhancement Program) for Strong Bonds is a standardized, evidence-based program conducted in a weekend residential retreat format with experiential exercises. The Army Chaplain Corps trains chaplains to facilitate the program. The manualized program uses methods from cognitive behavioral therapy and communication-oriented marital enhancement programs developed by Markman et al. at the Denver University Center for Marital and Family Studies. Topics include communication, conflict management, commitment, friendship, sensuality, problem-solving, and emotional supportiveness, among others.
  Arms: PREP only; PREP plus Mission Reconnect

SUMMARY:
An urgent and growing need exists for interventions that support the long-term adjustment and mental health needs of OIF/OEF veterans and their relationship partners after the return from deployment. This project will complete production of a multimedia intervention program for autonomous use, delivered by Internet and mobile app technology, that teaches couples selected mind/body interventions and massage techniques to promote stress reduction, compassion, resiliency and relationship re-integration. A four-armed randomized trial will evaluate mental health outcomes as a free-standing program and as complementary to a current standard of care structured group program.

DETAILED DESCRIPTION:
There is an urgent and growing need for mental health interventions supporting both short- and long-term reintegration of veterans of OIF and OEF into their communities and significant relationships. Innovative approaches are needed to support the well-being of veterans who may not access or be reached by formal services.

OBJECTIVES. This Phase II project will complete development and evaluation of a self-directed, home-based intervention to be used by OIF/OEF veterans and their loved ones to aid in the readjustment process. "Mission Reconnect" is an integrated program of (1) guided mind/body stress reduction and relaxation practices, (2) contemplative practices to engender and support appreciation, empathy and forgiveness for oneself and one's loved ones, and (3) video instruction in use of simple massage techniques with a partner for connection and stress reduction. Feasibility was established in Phase I with high user satisfaction and significant impact on measures of stress, depression, PTSD, and self-compassion, as well as qualitative data. In Phase II We will complete and evaluate the full program in a four-arm randomized controlled trial.

SPECIFIC AIMS. 1. Revise program content based on Phase I quantitative and qualitative data. 2. Film a diverse group of ten 10 veteran/partner dyads receiving and using revised material; use video footage for the final program. 3. Produce high quality audio and video components of the revised program. 4. Produce a multi-modal system for delivery of instructional components that leverages innovations in web-based and mobile device technologies to maximize access, utilization, and data collection. 5. Conduct an RCT with 160 dyads of OIF/OEF veterans and their chosen partners. 6. Evaluate impact of intervention on measures of stress, depression, PTSD symptoms, sleep quality, self-compassion, social support and relationship satisfaction. 7. Evaluate program utilization and satisfaction, massage effects, self-efficacy and satisfaction in users of the revised program.

IMPACT ON THE FIELD. Mission Reconnect offers a convenient, low cost resource helping users develop wellness skills to reduce current and future distress, enhance empathy and improve quality of life. The intervention can complement formal mental health services, or be used alone. This is a potential aid to the two million OIF/OEF veterans, their partners and families, as well as the 20 million living veterans of other eras, whose wounds of war can last for decades if unaddressed.

INNOVATION. The project leverages the dyadic relationship as a context for reciprocal and mutual use of complementary therapies for health promotion in both the veteran and partner. Project technology utilizes state of the art mobile app design, seamless integration across multiple devices, automated background data collection, and device-specific reminder alerts.

COMMERCIAL APPLICATION. The product will be marketed to family support programs of all branches of the military, VA system, and the private sector, including non-profit veterans' associations.

PRODUCT. Mission Reconnect is an integrated multimedia program deliverable over the Internet and mobile devices, and hard copy (DVD, CD, manual).

ELIGIBILITY:
Inclusion Criteria:

* Veteran of deployment in Operation Iraqi Freedom (OIF) or Operation Enduring Freedom (OEF)
* Partner or spouse of the veteran (veteran and partner/spouse must participate together in the project)

Exclusion Criteria:

* Couples are ineligible who have previously attended a PREP for Strong Bonds program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale (PSS-10) | Baseline, 2 months, 4 months
  Change from baseline to 2 months and 4 months
Change in Beck Depression Inventory (BDI) | Baseline, 2 months, 4 months
  Change from baseline to 2 months and 4 months
Change in Posttraumatic Checklist-Civilian (PCL-C) | Baseline, 2 months, 4 months
  Change from baseline to 2 months and 4 months
Change in The Self-Compassion Scale | Baseline, 2 months, 4 months
  Change from baseline to 2 months and 4 months
Change in Responses to Stressful Experiences Scale (RSES) | Baseline, 2 months, 4 months
  Change from baseline to 2 months and 4 months

SECONDARY OUTCOMES:
Change in Multidimensional Perceived Social Support Scale (MPSSS) | Baseline, 2 months, 4 months
  Change from baseline to 2 months and 4 months
Change in Pittsburgh Sleep Quality Index | Baseline, 2 months, 4 months
  Change from baseline to 2 months and 4 months
Change in Revised Dyadic Adjustment Scale (RDAS) | Baseline, 2 months, 4 months
  Change from baseline to 2 months and 4 months
Investigator-generated survey of use of stress reduction practices | Weekly for 8 weeks, then at 4 months
Investigator-generated survey on use of massage and massage effects | Weekly for 8 weeks
Investigator-generated survey on self-efficacy using massage, and satisfaction giving and receiving the use of massage | 2 months, 4 months
Investigator-generated ratings of program satisfaction | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: William B Collinge, PhD, MPH, Principal Investigator — Collinge and Associates, Inc.; Janet R Kahn, PhD, LMT, Principal Investigator — Peace Village Projects, Inc.

REFERENCES:
- [Background] Collinge W, Kahn J, Soltysik R. Promoting reintegration of National Guard veterans and their partners using a self-directed program of integrative therapies: a pilot study. Mil Med. 2012 Dec;177(12):1477-85. doi: 10.7205/milmed-d-12-00121. PMID 23397692
- [Derived] Kahn JR, Collinge W, Soltysik R. Post-9/11 Veterans and Their Partners Improve Mental Health Outcomes with a Self-directed Mobile and Web-based Wellness Training Program: A Randomized Controlled Trial. J Med Internet Res. 2016 Sep 27;18(9):e255. doi: 10.2196/jmir.5800. PMID 27678169
- See also: Website home of the Mission Reconnect Program — http://www.missionreconnect.com